CLINICAL TRIAL: NCT05346094
Title: A Multicenter Investigation of Cardiac Normal Values of Morphology, Function and Tissue Characteristics by Magnetic Resonance Imaging
Brief Title: Cardiac Normal Values Assessed by Magnetic Resonance Imaging
Status: Recruiting | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Minjie Lu, Chief Doctor, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: CMR_Normal
Record Dates: First submitted 2021-08-02; First posted 2022-04-26 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Healthy Participants; Reference Values
Keywords: reference values; morphology; function; tissue characterization; myocardial deformation; cardiocascular magnetic resonance imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study carried out a study enrolled healthy volunteers to comprehensively provide age and sex specific reference values of the normal cardiac structure and function of Chinese adults, using the steady-state free precession technique (SSFP) as well as reference values for novel cardiovascular magnetic resonance techniques including myocardial strian and tissue characterization.

DETAILED DESCRIPTION:
Cardiovascular magnetic resonance (CMR), as a non-invasive and radiation-free examination, can identify the structural and functional abnormalities of various cardiovascular diseases. It is the gold standard for cardiovascular structural and functional measurements, and recommended as a priority examination for cardiovascular diseases by guidelines of the American College of Cardiology (ACC/AHA) and the European College of Cardiology (ESC). The reference standard for cardiovascular structure and function of normal people is the basis for cardiovascular disease study, and plays a vital role in diagnosis, differential diagnosis, and prognosis evaluation. CMR parameters have been shown to provide significant information for the general population and have always been important biomarkers for morbidity and mortality in patients with cardiac pathologies. Although there are relevant reference standards for normal values in the world, there is no standard for normal values of large samples of Chinese people. In addition, most of the normal values are limited to traditional parameters of cardiac structure and function, and there is no normal value standard for novel parameters including myocardial strain and tissue characteristics. Therefore, on the basis of previous works, our group planned to create a cardiovascular MRI reference value database of normal Chinese people through retrospective and prospective recruitment, which will lay a foundation for the early identification and prognosis assessment of cardiovascular diseases, and promote the progress of systematic cardiovascular magnetic resonance studies.

ELIGIBILITY:
Inclusion Criteria:

Subjects without cardiovascular disease, cardiovascular related symptoms and risk factors judged by combining clinical manifestations, non-invasive imaging and laboratory examination

Exclusion Criteria:

* Subjects clinically screened or previously diagnosed with cardiovascular disease and risk factors
* Subjects with serious non-cardiovascular diseases
* Subjects with poor quality of magnetic resonance imaging
* Subjects refused to participate in the study
* Subjects with contraindications to MRI

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy subjects without cardiovascular disease, cardiovascular related symptoms and risk factors judged by combining clinical manifestations, non-invasive imaging and laboratory examination
Sampling Method: Probability Sample
Enrollment: 938 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Normal values of left and right structures and cardiac function | 5 years
  Create a database for normal values of left and right structures and cardiac function
Normal values of novel cardiovascular magnetic resonance parameters | 5 years
  Create a database for normal values of novel cardiovascular magnetic resonance parameters

CONTACTS AND LOCATIONS:
Overall Officials: Minjie Lu, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] von Knobelsdorff-Brenkenhoff F, Pilz G, Schulz-Menger J. Representation of cardiovascular magnetic resonance in the AHA / ACC guidelines. J Cardiovasc Magn Reson. 2017 Sep 25;19(1):70. doi: 10.1186/s12968-017-0385-z. PMID 28942735
- [Result] von Knobelsdorff-Brenkenhoff F, Schulz-Menger J. Role of cardiovascular magnetic resonance in the guidelines of the European Society of Cardiology. J Cardiovasc Magn Reson. 2016 Jan 22;18:6. doi: 10.1186/s12968-016-0225-6. PMID 26800662
- [Result] Zhou D, Xu J, Zhao S, Lu M. CMR publications from China of the last more than 30 years. Int J Cardiovasc Imaging. 2020 Sep;36(9):1737-1747. doi: 10.1007/s10554-020-01873-x. Epub 2020 May 11. PMID 32394180
- [Result] Bruder O, Wagner A, Lombardi M, Schwitter J, van Rossum A, Pilz G, Nothnagel D, Steen H, Petersen S, Nagel E, Prasad S, Schumm J, Greulich S, Cagnolo A, Monney P, Deluigi CC, Dill T, Frank H, Sabin G, Schneider S, Mahrholdt H. European Cardiovascular Magnetic Resonance (EuroCMR) registry--multi national results from 57 centers in 15 countries. J Cardiovasc Magn Reson. 2013 Jan 18;15(1):9. doi: 10.1186/1532-429X-15-9. PMID 23331632
- [Result] Klinke V, Muzzarelli S, Lauriers N, Locca D, Vincenti G, Monney P, Lu C, Nothnagel D, Pilz G, Lombardi M, van Rossum AC, Wagner A, Bruder O, Mahrholdt H, Schwitter J. Quality assessment of cardiovascular magnetic resonance in the setting of the European CMR registry: description and validation of standardized criteria. J Cardiovasc Magn Reson. 2013 Jun 20;15(1):55. doi: 10.1186/1532-429X-15-55. PMID 23787094
- [Result] Bruder O, Schneider S, Nothnagel D, Pilz G, Lombardi M, Sinha A, Wagner A, Dill T, Frank H, van Rossum A, Schwitter J, Nagel E, Senges J, Sabin G, Sechtem U, Mahrholdt H. Acute adverse reactions to gadolinium-based contrast agents in CMR: multicenter experience with 17,767 patients from the EuroCMR Registry. JACC Cardiovasc Imaging. 2011 Nov;4(11):1171-6. doi: 10.1016/j.jcmg.2011.06.019. PMID 22093267
- [Result] Global Cardiovascular Magnetic Resonance Registry (GCMR) Investigators; Kwong RY, Petersen SE, Schulz-Menger J, Arai AE, Bingham SE, Chen Y, Choi YL, Cury RC, Ferreira VM, Flamm SD, Steel K, Bandettini WP, Martin ET, Nallamshetty L, Neubauer S, Raman SV, Schelbert EB, Valeti US, Cao JJ, Reichek N, Young AA, Fexon L, Pivovarov M, Ferrari VA, Simonetti OP. The global cardiovascular magnetic resonance registry (GCMR) of the society for cardiovascular magnetic resonance (SCMR): its goals, rationale, data infrastructure, and current developments. J Cardiovasc Magn Reson. 2017 Jan 20;19(1):23. doi: 10.1186/s12968-016-0321-7. PMID 28187739
- [Result] Esposito A, Gallone G, Palmisano A, Marchitelli L, Catapano F, Francone M. The current landscape of imaging recommendations in cardiovascular clinical guidelines: toward an imaging-guided precision medicine. Radiol Med. 2020 Nov;125(11):1013-1023. doi: 10.1007/s11547-020-01286-9. Epub 2020 Sep 22. PMID 32964326